CLINICAL TRIAL: NCT03198494
Title: Low Frequency Acoustic Stimulation During Sleep for Seizure Suppression
Brief Title: Acoustic Stimulation for Seizure Suppression
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 17-00698
Record Dates: First submitted 2017-06-16; First posted 2017-06-26 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Epilepsy
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Acoustic 1Hz Stimulation (Experimental): 1 Hz acoustic stimulation applied via headphones and downloadable phone application during sleep every night.
  Interventions: Other: Acoustic 1Hz Stimulation
- Sham Background Noise (Sham Comparator): Background noise applied via headphones and downloadable phone application during sleep every night.
  Interventions: Other: Sham Background Noise
- Baseline Seizure Monitoring (No Intervention): No use of sound system; Patients record seizures in a diary.

INTERVENTIONS:
Other: Acoustic 1Hz Stimulation — 1Hz acoustic pulses delivered during sleep via headphones
  Arms: Acoustic 1Hz Stimulation
Other: Sham Background Noise — Background Noise used as a control
  Arms: Sham Background Noise

SUMMARY:
The objective of this study is to test the feasibility and physiological effect of low-frequency (1 Hz) acoustic stimulation delivered during nocturnal NREM sleep in epilepsy patients. The long-term goal is to develop this protocol for daily, long-term use in a home setting, for nocturnal seizure and IED suppression

DETAILED DESCRIPTION:
1. To test the feasibility of wearing an earphone system delivering acoustic stimulation during a night of sleep in adult epilepsy patients monitored in an inpatient unit.
2. To determine the acute physiological effects of low-frequency acoustic stimulation on interictal epileptiform discharge (IED) frequency during NREM sleep in adult patients with epilepsy in an ambulatory setting.
3. To determine the feasibility of applying low-frequency acoustic stimulation in a long-term home setting in adult epilepsy patients with frequent nocturnal seizures.

ELIGIBILITY:
Inclusion Criteria:

* 18-60 years old
* Able to provide informed consent
* MOCA ≥26
* Fluent in English
* Frequent nocturnal IEDs (≥ 10% of the sleep record)
* Monitored on the adult epilepsy monitoring unit (EMU, for Aim 1 only) Additional inclusion criteria for Aim 3
* Frequent nocturnal seizures (≥1 per week)

Exclusion Criteria:

* Hearing impairment
* Diagnosis of a sleep disorder (sleep apnea, periodic limb movements of sleep, or other medical conditions with frequent arousals)
* Psychoactive medication use (other than AEDs, for example SSRIs, antipsychotics, BDZ, or stimulants)
* Seizures ≤ 24 hours prior to study.
* Alcohol or recreational drug use in the 24 hours prior to the study
* BMI ≥ 30
* MOCA <26
* History of recent travel across time zones within the 1 month prior to study activities
* Shift work for 1 month prior to study activities Additional Exclusion Criteria for Aim 3
* No medication changes at least 1 month before study, and during 3 months of study activities

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2017-08-17 (Actual); Primary Completion 2028-11-21 (Estimated); Study Completion 2028-11-21 (Estimated)

PRIMARY OUTCOMES:
Successful System Training | 72 hours
  Assessment of how well participants learn to use stimulation smart-phone application and headphones, defined as the percentage of subjects with correctly maintained earphones during the first four hours of nocturnal sleep in the first days of use.
Interictal Discharge frequency | 72 hours
  IED frequency during nighttime sleep as measured by a 72 hour ambulatory EEG
System Adherence | 2 months
  Percentage of nights during which patients were compliant with the acoustic stimulation device during two months of home use (1 month control acoustic condition, 1 month 1Hz stimulation) determined weekly by patient self-report

SECONDARY OUTCOMES:
System Use effect on Features of Sleep | 72 hours
  Effect of system use on sleep features, including time spent in each stage of sleep, delta and spindle power and spatial distribution gather from EEG.
Seizure Control | 3 months
  Seizure frequency during control and treatment months gathered from seizure diary and IED frequency gathered from EEG (1 month baseline, 1 month sham stimulation, 1 month 1Hz stimulation).

CONTACTS AND LOCATIONS:
Overall Officials: Anli Liu, Principal Investigator — NYU Langone Health
Locations (1):
- New York University School of Medicine, New York, New York, United States